CLINICAL TRIAL: NCT07030621
Title: Efficacy of Semaglutide in Improving Neurological Outcomes After Endovascular Thrombectomy for Acute Ischemic Stroke: A Randomized Double-Blind Controlled Trial
Acronym: STARS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-175
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Ischemic Stroke
Keywords: endovascular thrombectomy; semaglutide
MeSH Terms: conditions — Ischemic Stroke | interventions — semaglutide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide group (Experimental): The patients will receive a subcutaneous injection of 0.5 mg semaglutide into the abdomen during endovascular thrombectomy
  Interventions: Drug: Semaglutide 0.5 mg
- placebo group (Placebo Comparator): The patients in the control group will receive a similar-looking Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Semaglutide 0.5 mg — Semaglutide is a glucagon-like peptide-1 receptor agonist (GLP-1 RA) analog, which has been found to have neuroprotective effects.
  Arms: semaglutide group
Drug: Normal Saline — Normal saline is the placebo drug.
  Arms: placebo group

SUMMARY:
The trial will be a randomized, double-blind, controlled, single-center trial. The purpose of this trial is to determine the efficacy and safety of semaglutide in improving neurological outcomes after endovascular thrombectomy for acute ischemic stroke. The patients in the treatment group will receive a subcutaneous injection of 0.5 mg semaglutide into the abdomen during endovascular thrombectomy. The patients in the control group will receive a similar-looking placebo. Patients will be randomized to the treatment or control group by the pharmacy, eliminating the selection bias. The patient and evaluator will be blind to the allocation of patients, further minimizing the bias.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a condition associated with high rates of disability and mortality worldwide, and its incidence continues to rise in our country. Endovascular thrombectomy (EVT), a major advance in stroke treatment in recent years, has gained widespread clinical application and become a standard treatment for AIS caused by large-vessel occlusion. EVT significantly improves neurological functional outcomes. However, in clinical practice, despite successful recanalization of the occluded artery, nearly half of patients do not achieve a favorable prognosis. There is a compelling need to identify novel neuroprotective strategies to enhance the effectiveness of EVT and improve patient quality of life.

Recent evidence indicates that semaglutide reduces neuroinflammation and is associated with a decreased risk of stroke and fewer neurological complications in patients with diabetes. We anticipate that this trial will provide valuable insights into the potential role of semaglutide as a neuroprotective agent in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or imaging diagnosis of acute ischemic stroke within 24 hours after onset;
2. Scheduled for endovascular thrombectomy;
3. Age ≥18 years;
4. Pre-stroke modified Rankin Scale (mRS) score ≤1;
5. Informed consent voluntarily signed by the patient or legal representative.

Exclusion Criteria:

1. Preoperative imaging diagnosis of intracranial hemorrhage, or history of intracranial hemorrhage within 3 months prior to surgery;
2. Contraindications for endovascular thrombectomy;
3. Recent history of ischemic stroke;
4. Fasting blood glucose <3.9 mmol/L;
5. ASA classification of IV-V;
6. Severe organic heart disease or severe arrhythmia;
7. Pregnant or lactating women;
8. Contraindications to semaglutide or allergy to semaglutide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
mRS at 90-days | 90 days postoperatively
  The primary endpoint is the degree of disability or dependence at 90 days as assessed by the mRS shift. A global measure of disability, the mRS comprises of seven grades ranging from 0 (no symptoms) to 6 (death). 0-2 points: indicating good neurological function recovery in patients; 3-6 points: indicating poor neurological function recovery in patients.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) at 24 hours and 7-days | A decrease of ≥8 points in the NIHSS score from baseline to 24 hours and 7 days postoperatively, or a score of 0 to 1, indicates neurological improvement; an increase of ≥4 points indicates neurological deterioration.
  NIHSS at 24 hours and 7-days will be recorded based on the patient's neurologic status by a health care professional to assess stroke severity post-procedure.
Infarct volume after 72 hours of treatment | 72 hours postoperatively
  assessed by magnetic resonance imaging brain scan
the incidence of surgical complications within 90 days postoperatively | within 90 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Casares N, Gonzalez-Gonzalez G, de la Cruz-Cosme C, Garzon-Maldonado FJ, de Rojas-Leal C, Ariza MJ, Narvaez M, Barbancho MA, Garcia-Arnes JA, Tinahones FJ. Effects of GLP-1 receptor agonists on neurological complications of diabetes. Rev Endocr Metab Disord. 2023 Aug;24(4):655-672. doi: 10.1007/s11154-023-09807-3. Epub 2023 May 26. PMID 37231200
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Cui QN, Stein LM, Fortin SM, Hayes MR. The role of glia in the physiology and pharmacology of glucagon-like peptide-1: implications for obesity, diabetes, neurodegeneration and glaucoma. Br J Pharmacol. 2022 Feb;179(4):715-726. doi: 10.1111/bph.15683. Epub 2021 Nov 23. PMID 34519040
- [Background] Li Y, Fan Q, Pang R, Cai L, Qi J, Chen W, Zhang Y, Chen C, Yu W, Li P. Semaglultide targets Spp1+ microglia/macrophage to attenuate neuroinflammation following perioperative stroke. J Neuroinflammation. 2025 May 27;22(1):143. doi: 10.1186/s12974-025-03465-9. PMID 40426210
- [Background] Candelario-Jalil E, Dijkhuizen RM, Magnus T. Neuroinflammation, Stroke, Blood-Brain Barrier Dysfunction, and Imaging Modalities. Stroke. 2022 May;53(5):1473-1486. doi: 10.1161/STROKEAHA.122.036946. Epub 2022 Apr 7. PMID 35387495
- [Background] DeLong JH, Ohashi SN, O'Connor KC, Sansing LH. Inflammatory Responses After Ischemic Stroke. Semin Immunopathol. 2022 Sep;44(5):625-648. doi: 10.1007/s00281-022-00943-7. Epub 2022 Jun 29. PMID 35767089
- [Background] Nie X, Leng X, Miao Z, Fisher M, Liu L. Clinically Ineffective Reperfusion After Endovascular Therapy in Acute Ischemic Stroke. Stroke. 2023 Mar;54(3):873-881. doi: 10.1161/STROKEAHA.122.038466. Epub 2022 Dec 7. PMID 36475464
- [Background] Yoshimura S, Sakai N, Yamagami H, Uchida K, Beppu M, Toyoda K, Matsumaru Y, Matsumoto Y, Kimura K, Takeuchi M, Yazawa Y, Kimura N, Shigeta K, Imamura H, Suzuki I, Enomoto Y, Tokunaga S, Morita K, Sakakibara F, Kinjo N, Saito T, Ishikura R, Inoue M, Morimoto T. Endovascular Therapy for Acute Stroke with a Large Ischemic Region. N Engl J Med. 2022 Apr 7;386(14):1303-1313. doi: 10.1056/NEJMoa2118191. Epub 2022 Feb 9. PMID 35138767
- [Background] Lansberg MG, Schrooten M, Bluhmki E, Thijs VN, Saver JL. Treatment time-specific number needed to treat estimates for tissue plasminogen activator therapy in acute stroke based on shifts over the entire range of the modified Rankin Scale. Stroke. 2009 Jun;40(6):2079-84. doi: 10.1161/STROKEAHA.108.540708. Epub 2009 Apr 16. PMID 19372447
- [Background] Powers WJ. Acute Ischemic Stroke. N Engl J Med. 2020 Jul 16;383(3):252-260. doi: 10.1056/NEJMcp1917030. No abstract available. PMID 32668115
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721